CLINICAL TRIAL: NCT02847780
Title: Assessment of Vocal Cord Movement After Thyroid Surgery Using C-MAC Video-laryngoscope and Airway Ultrasound.
Brief Title: Comparison of Two Technique for Assessment of Vocal Cord Movement by C-Mac Videolaryngoscope vs Airway Ultrasound.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Amit Kumar Mittal, Consultant in-charge, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 505/AN/AKM-03
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2017-04

CONDITIONS: Objective Vocal Cord Movement Assessment by C-Mac Videolaryngoscope Vs Airway Ultrasound in Ca Thyroid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C-Mac video laryngoscope. (Active Comparator): Active Comparator: C-Mac Videolaryngoscope for vocal cord movement assessment.
  Interventions: Device: Active Comparator :C-Mac Videolaryngoscope; Device: Experimental: Airway ultrasound,
- Airway Ultrasound (Experimental): Experimental: Airway Ultrasound for vocal cord movement assessment.
  Interventions: Device: Active Comparator :C-Mac Videolaryngoscope; Device: Experimental: Airway ultrasound,

INTERVENTIONS:
Device: Active Comparator :C-Mac Videolaryngoscope — Real time assessment of Glottic aperture at the time of extubation by videolaryngoscope
Device: Experimental: Airway ultrasound, — Airway ultrasound using portable ultrasound machine to assess vocal cords movement.

SUMMARY:
This study is planned to compare C-Mac video-laryngoscope and airway ultrasound as two novel techniques (causing least discomfort to the patients) for the detection of impaired vocal-cord movement after thyroid surgery.

DETAILED DESCRIPTION:
In this prospective study 100 patients posted for Thyroid surgery will be included, after explaining the procedure and written informed consent, all included patients in the study will be assessed for vocal cord mobility by C-Mac video laryngoscope (manufactured by KARL STORZ Video Laryngoscopes) followed by airway ultrasonography (USG). Linear transducer (7.5 MHz) will be used for scanning the airway placed at the level of thyroid cartilage with 10-15 degree cephalad tilt so to get proper acoustic window and for optimal visualization of laryngeal structures. C-Mac video laryngoscope will be required for virtual visualization of glottis apertures and vocal cord movement. All patients will be scanned pre-operatively by indirect laryngoscopy to see vocal cord mobility as a reference value. Immediately after extubation the patient will be scanned for vocal cord mobility by videolaryngoscope by first examiner, After oxygenation and stabilization of haemodynamic, ultrasound of airway will be performed to study the vocal cord movement by the other examiner (blinded to the laryngoscopy finding).Visibility of false vocal cords, true vocal cords and arytenoids will be given one point each for one side, maximal score will be 6. According to points the acoustic window scoring for glottis aperture will be graded as fair (score1-2), good(score3-4) and very good(score5-6) Findings of both the examiners will be collected by the primary investigator for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient's undergoing thyroid and parathyroid surgery.

Exclusion Criteria:

* patients not extubated.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
• To determine objective vocal cord mobility by the video laryngoscope and airway ultrasound | At time of extubation.
  patients vocal cords will be assessed by videolaryngoscope at time of extubation then the cords will be again assessed by airway ultrasound.

SECONDARY OUTCOMES:
• To ascertain whether airway ultrasound can be used as a reliable alternative to assess post-operative vocal cord mobility | After extubation and before dressing.
  After extubation with aseptic precaution patient's airway will be scanned for vocal cord movement assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Amit kr Mittal, M.D, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre, Rohini; New Delhi: India 110085.
Locations (1):
- Rajiv Gandhi Cancer Institute & Research center, Rohini, New Delhi, India

IPD SHARING:
Plan to Share IPD: No